CLINICAL TRIAL: NCT05430659
Title: Intraoperative Estimated Blood Loss, Blood Transfusion, and Postoperative Clinical Outcomes in Patients Undergoing Non Cardiac Surgery, Siriraj Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Principal Investigator, Siriraj Hospital
Other Study IDs: 333/2565
Record Dates: First submitted 2022-06-15; First posted 2022-06-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: General Surgery; Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EBL equal or more than 500 ml: The intraoperative estimated blood loss equal or more than 500 ml
  Interventions: Other: observational study
- EBL less than 500 ml: The intraoperative estimated blood loss less than 500 ml
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Retrospective observational study

SUMMARY:
After review literature, Siriraj hospital has not unanimous protocol to guide proper preoperative anemia and blood transfusion. This retrospective study will review non-cardiac surgery cases and collect data such as demographic data, surgical procedures, anesthetic techniques, preoperative hemoglobin level, intraoperative estimate blood loss, blood transfusion, and post operative complication in Siriraj hospital which has many patients undergo various operations. This study can be model to develop preoperative anemia management guideline in Siriraj Preanesthesia Assessment Center (SIPAC), Siriraj hospital and reduce risk and adverse outcomes after blood transfusion in the future.

DETAILED DESCRIPTION:
One of the worldwide health problems that covers more than a quarter of the population is anemia. The World Health Organization (WHO) recommendations use of hemoglobin concentration for diagnosing anemia as hemoglobin (Hb) level <12 g/dL and < 13 g/dL for women and men, respectively. The most of anemic patients caused by iron deficiency anemia (IDA), followed by the anemia of chronic disease (ACD).

Iron deficiency anemia often result from malnutrition status, acute or chronic blood loss such as perioperative blood loss. Chronic kidney disease is the primary cause of anemia of chronic disease, followed by acute or chronic inflammatory conditions, or in patients with malignancies.Currently, there are lack of preoperative evaluation, diagnostic methods, and adequate treatments for anemia before attaining elective non cardiac surgery. Baron et al retrospective study the European Surgical Outcome included 39,309 patients from 28 European countries. The prevalence of anemic patients was about 26.5% in women and 31.1% in men. The higher rate of prolonged hospital administration (P = .0001) and transferred to intensive care unit (P = .001) in moderate to severe anemic patients. Moreover, anemic patients who undergone cardiac surgery and non-cardiac surgery showed a higher mortality than nonanemic patients.

Preoperative hemoglobin level was used with other factors such as demographic data, surgical procedures, and anesthetic technique to increase predictive accuracy of perioperative blood transfusion. The mortality rate raised in anemic patients who received blood transfusion in perioperative period. Criteria for blood transfusion had various factors. The important factor which usually used is hemoglobin level: Liberal strategy suggested starting blood transfusion when Hb level below 9-10 g/dL, another method was Restrictive strategy that starting blood transfusion if Hb level below 7-8 g/dL. In addition, the hemoglobin threshold cut-off point level often differed due to the objective for each study.Althrough many organizations tried to develop standard protocol for blood transfusion, the universal transfusion threshold level cloud not properly use for all patients.Blood transfusion remained the cornerstone of the treatment of anemia but intraoperative period inappropriately transfused blood component causing risk of post operative complication, 30-days mortality, increasing length of hospital stay, and transferring to intensive care unit.

Moreover, The National Blood Authority studied about types of operation and operation at risk for blood transfusion that had operative time more than 2 hours and estimated blood loss more than 500 ml, needed to receive blood transfusion before surgery. The American College of Cardiology had found various factors affecting peri-operative blood transfusion risk but they were not practical to use in real-life practice.

After review literature, Siriraj hospital has not unanimous protocol to guide proper preoperative anemia and blood transfusion. This retrospective study will review non-cardiac surgery cases and collect data such as demographic data, surgical procedures, anesthetic techniques, preoperative hemoglobin level, intraoperative estimate blood loss, blood transfusion, and post operative complication in Siriraj hospital which has many patients undergo various operations. This study can be model to develop preoperative anemia management guideline in Siriraj Preanesthesia Assessment Center (SIPAC), Siriraj hospital and reduce risk and adverse outcomes after blood transfusion in the future.

ELIGIBILITY:
Inclusion criteria:

Patients undergoing surgical procedures consist of head/neck surgery, general surgery, urologic surgery, vascular surgery, neurologic surgery, orthopedic surgery, otolaryngologic surgery and gynecologic surgery.

Exclusion Criteria:

Patients don't have target data or losing of interesting document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical procedures consist of head/neck surgery, general surgery, urologic surgery, vascular surgery, neurologic surgery, orthopedic surgery, otolaryngologic surgery and gynecologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1268 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Operation with intraoperative blood loss of more than 500 ml | Day of surgery
  Operation with intraoperative blood loss of more than 500 ml

SECONDARY OUTCOMES:
Risks associated with intraoperative blood loss of more than 500 ml | Day of surgery
  Risks associated with intraoperative blood loss of more than 500 ml

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided